CLINICAL TRIAL: NCT00132691
Title: Multicenter Uveitis Steroid Treatment (MUST) Trial
Acronym: MUST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JHSPH Center for Clinical Trials (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-106; U10EY014660 (NIH); 1U10EY014660-2; ISRCTN15396562; NCT00269698 (obsolete NCT alias)
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-10

CONDITIONS: Uveitis
Keywords: uveitis; non-infectious intermediate uveitis; non-infectious posterior uveitis; non-infectious panuveitis
MeSH Terms: conditions — Uveitis | interventions — Adrenal Cortex Hormones; Immunosuppressive Agents; Health Services Needs and Demand; Alkylating Agents; Cyclophosphamide; Azathioprine; Chlorambucil; Methotrexate; Mycophenolic Acid; Cyclosporine; Tacrolimus; Biological Products; Infliximab; Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Immunosuppressant medication implant
  Interventions: Drug: fluocinolone acetonide intraocular implant
- 2 (Active Comparator): Systemic corticosteroids with immunosuppressant drugs as needed
  Interventions: Drug: oral corticosteroid with immunosuppressive agents as needed

INTERVENTIONS:
Drug: fluocinolone acetonide intraocular implant — RETISERT™ (fluocinolone acetonide intravitreal implant) 0.59 mg is a sterile implant designed to release fluocinolone acetonide locally to the posterior segment of the eye at a nominal initial rate of 0.6 μg/day, decreasing over the first month to a steady state between 0.3-0.4 μg/day over approximately 30 months.
  Other Names: NDC 24208-416-01
  Arms: 1
Drug: oral corticosteroid with immunosuppressive agents as needed — Prednisone
  Other Names: Permitted immunosuppressive agents:; - Alkylating agents; cyclophosphamide (Cytoxan); chlorambacil; - Antimetabolities; azathioprine (Imuran); azathioprine chlorambucil (Leukeran); methotrexate (Rheumatrex and others); mycophenolate mofetil (Cellcept); - T-cell inhibitors; cyclosporine (Neoral, Sandimmune and other trade names); tacrolimus; - Biologics; infliximab; daclizumab; other biologics
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effectiveness of standardized systemic therapy versus fluocinolone acetonide implant therapy for the treatment of severe cases of non-infectious intermediate uveitis, posterior uveitis, or panuveitis.

DETAILED DESCRIPTION:
The MUST trial is a randomized controlled clinical trial comparing two treatments for patients with vision-threatening non-infectious intermediate uveitis, posterior uveitis, or panuveitis:

* local therapy with fluocinolone acetonide intraocular implant in affected eyes; versus
* standard therapy: systemic corticosteroid therapy supplemented, when indicated, by corticosteroid-sparing potent immuno-modulator therapy.

Study ophthalmologists, clinic coordinators, and patients will not be masked to treatment assignment. Masking will be applied to the determination of visual function at baseline, the six month visit, and thereafter . Patients will be followed until death, participant withdrawal, or a common study closeout. Patients will be seen at baseline, one month after randomization, three months after randomization, and every three months thereafter for data collection. Both ophthalmological and medical data will be collected to evaluate the outcomes of treatment of the uveitis, complications of the uveitis, and complications from therapy itself. Selected laboratory data related to the complications from systemic corticosteroid therapy will be collected.

The planned sample size of 250 patients, 125 per treatment group, is expected to give sufficient power to detect clinically important differences in visual acuity outcomes. Patients meeting the eligibility criteria detailed above will be enrolled at approximately 23 clinical centers in the United States, Australia and UK. Patients will be randomized on a 1:1 basis to one of the two treatment groups.

The MUST Research Group received additional funding at the completion of the MUST Trial to continue following patients enrolled in the study for an additional 7 years in the MUST Trial Follow-up Study (MUST FS). Since uveitis is often a chronic condition requiring long-term treatment, the objectives of the MUST FS are to evaluate outcomes of the two treatments over a longer period time. The outcomes specified for MUST FS are the same as those specified for the MUST Trial: visual acuity, ocular and systemic side effects of treatment, quality of life, and control of ocular inflammation. The primary analyses will be to compare outcomes between the original randomization groups, i.e., intention-to-treat. Secondary analyses will be based on treatment received. Study visits will be conducted every 6 months in MUST FS as opposed to every 3 months in the MUST Trial. Two analyses are planned for public release, one at 4.5 years and one after 7 years of follow-up. The Data Safety Monitoring Board reviewed and approved the analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 years or older
* Best-corrected visual acuity of hand motions or better in at least one eye with uveitis
* Intraocular pressure 24 mm Hg or less in all eyes with uveitis

Exclusion Criteria:

* Inadequately controlled diabetes
* Uncontrolled glaucoma
* Advanced glaucomatous optic nerve injury
* A history of scleritis; presence of an ocular toxoplasmosis scar.
* HIV infection or other immunodeficiency disease for which corticosteroid therapy would be contraindicated according to best medical judgment

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2005-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Jabs, MD, MBA, Study Chair — Icahn School of Medicine at Mount Sinai; John Kempen, MD, PhD, Study Chair — Scheie Eye Center, University of Pennsylvania; Janet T Holbrook, PhD, MPH, Study Director — Director of Coordinating Cener, Johns Hopkins Bloomberg School of Public Health; Michael Altaweel, MD, Study Director — Director of Fundus Photography Reading Center, University of Wisconsin at Madison
Locations (23):
- United States (21):
  - Jacobs Retina Center, UCSD, La Jolla, California
  - Doheny Eye Institute, USC, Los Angeles, California
  - Jules Stein Eye Institute, UCLA, Los Angeles, California
  - Proctor Foundation, UCSF, San Francisco, California
  - Anne Bates Leach Eye Hospital, University of Miami Miller School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago Eye Center, Chicago, Illinois
  - Wilmer Eye Institute, Johns Hopkins University, Baltimore, Maryland
  - National Eye Institute, NIH, Bethesda, Maryland
  - Massachusetts Eye Research & Surgery Institute, Cambridge, Massachusetts
  - Kellogg Eye Center, University of Michigan, Ann Arbor, Michigan
  - Barnes Retina Institute, St Louis, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - Duke Eye Center, Duke University, Durham, North Carolina
  - Scheie Eye Institute, University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Retina Associates, Dallas, Texas
  - Vitreoretinal Consultants, Houston, Texas
  - John A. Moran Eye Center, University of Utah, Salt Lake City, Utah
  - Virginia Eye Consultants, Norfolk, Virginia
- Royal Victoria Eye & Ear Hospital, East Melbourne, Australia
- United Kingdom Institute of Ophthalmology, London, United Kingdom

REFERENCES:
- [Result] Multicenter Uveitis Steroid Treatment (MUST) Trial Research Group; Kempen JH, Altaweel MM, Holbrook JT, Jabs DA, Louis TA, Sugar EA, Thorne JE. Randomized comparison of systemic anti-inflammatory therapy versus fluocinolone acetonide implant for intermediate, posterior, and panuveitis: the multicenter uveitis steroid treatment trial. Ophthalmology. 2011 Oct;118(10):1916-26. doi: 10.1016/j.ophtha.2011.07.027. Epub 2011 Aug 15. PMID 21840602
- [Derived] Tomkins-Netzer O, Lightman SL, Burke AE, Sugar EA, Lim LL, Jaffe GJ, Altaweel MM, Kempen JH, Holbrook JT, Jabs DA; Multicenter Steroid Treatment Trial and Follow-up Study Research Group. Seven-Year Outcomes of Uveitic Macular Edema: The Multicenter Uveitis Steroid Treatment Trial and Follow-up Study Results. Ophthalmology. 2021 May;128(5):719-728. doi: 10.1016/j.ophtha.2020.08.035. Epub 2020 Sep 10. PMID 32918964
- [Derived] Writing Committee for the Multicenter Uveitis Steroid Treatment (MUST) Trial and Follow-up Study Research Group; Kempen JH, Altaweel MM, Holbrook JT, Sugar EA, Thorne JE, Jabs DA. Association Between Long-Lasting Intravitreous Fluocinolone Acetonide Implant vs Systemic Anti-inflammatory Therapy and Visual Acuity at 7 Years Among Patients With Intermediate, Posterior, or Panuveitis. JAMA. 2017 May 16;317(19):1993-2005. doi: 10.1001/jama.2017.5103. PMID 28477440
- [Derived] Yu T, Holbrook JT, Thorne JE, Puhan MA. Using a patient-centered approach to benefit-harm assessment in treatment decision-making: a case study in uveitis. Pharmacoepidemiol Drug Saf. 2016 Apr;25(4):363-71. doi: 10.1002/pds.3959. Epub 2016 Jan 22. PMID 26798977
- [Derived] Yu T, Holbrook JT, Thorne JE, Flynn TN, Van Natta ML, Puhan MA. Outcome Preferences in Patients With Noninfectious Uveitis: Results of a Best-Worst Scaling Study. Invest Ophthalmol Vis Sci. 2015 Oct;56(11):6864-72. doi: 10.1167/iovs.15-16705. PMID 26501236
- [Derived] Drye LT, Casper AS, Sternberg AL, Holbrook JT, Jenkins G, Meinert CL. The transitioning from trials to extended follow-up studies. Clin Trials. 2014 Dec;11(6):635-47. doi: 10.1177/1740774514547396. Epub 2014 Aug 12. PMID 25115882
- [Derived] Domalpally A, Altaweel MM, Kempen JH, Myers D, Davis JL, Foster CS, Latkany P, Srivastava SK, Stawell RJ, Holbrook JT; MUST Trial Research Group. Optical coherence tomography evaluation in the Multicenter Uveitis Steroid Treatment (MUST) trial. Ocul Immunol Inflamm. 2012 Dec;20(6):443-7. doi: 10.3109/09273948.2012.719258. Epub 2012 Nov 19. PMID 23163490
- [Derived] Sen HN, Drye LT, Goldstein DA, Larson TA, Merrill PT, Pavan PR, Sheppard JD, Burke A, Srivastava SK, Jabs DA; Multicenter Uveitis Steroid Treatment (MUST) Trial Research Group. Hypotony in patients with uveitis: The Multicenter Uveitis Steroid Treatment (MUST) Trial. Ocul Immunol Inflamm. 2012 Apr;20(2):104-12. doi: 10.3109/09273948.2011.647228. PMID 22409563
- [Derived] Frick KD, Drye LT, Kempen JH, Dunn JP, Holland GN, Latkany P, Rao NA, Sen HN, Sugar EA, Thorne JE, Wang RC, Holbrook JT; Multicenter Uveitis Steroid Treatment-MUST Trial Research Group. Associations among visual acuity and vision- and health-related quality of life among patients in the multicenter uveitis steroid treatment trial. Invest Ophthalmol Vis Sci. 2012 Mar 9;53(3):1169-76. doi: 10.1167/iovs.11-8259. Print 2012 Mar. PMID 22247489
- [Derived] Sugar EA, Jabs DA, Altaweel MM, Lightman S, Acharya N, Vitale AT, Thorne JE; Multicenter Uveitis Steroid Treatment (MUST) Trial Research Group. Identifying a clinically meaningful threshold for change in uveitic macular edema evaluated by optical coherence tomography. Am J Ophthalmol. 2011 Dec;152(6):1044-1052.e5. doi: 10.1016/j.ajo.2011.05.028. Epub 2011 Sep 8. PMID 21861971
- [Derived] Madow B, Galor A, Feuer WJ, Altaweel MM, Davis JL. Validation of a photographic vitreous haze grading technique for clinical trials in uveitis. Am J Ophthalmol. 2011 Aug;152(2):170-176.e1. doi: 10.1016/j.ajo.2011.01.058. Epub 2011 Jun 8. PMID 21652026
- See also: MUST, JHU, Center for Clinical Trials — http://www.musttrial.org/
- See also: ISRCTN15396562 — http://www.controlled-trials.com/ISRCTN15396562/multicenter+uveitis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were enrolled at 23 uveitis centers in the US, the United Kingdom and Australia from 6 December 2005 to 9 December 2008.
Pre-assignment Details: 579 patients were assessed for initial eligibility (e.g. through chart review). Patients who were potentially eligible and interested in joining the trial signed an informed consent and underwent a baseline visit to confirm eligibility. Eligible patients (255) were randomly assigned to systemic treatment or implant treatment.
Groups:
- Flucinolone Acetonide Intraocular Implant: Local therapy with fluocinolone acetonide 0.59 mg implant (Retisert; Bausch & Lomb Inc.) in each eye with uveitis of sufficient severity to justify treatment with systemic corticosteroids
- Standard Systemic Treatment: Systemic corticosteroid therapy with immunosuppression as indicated
Period: Overall Study
Arm/Group | Flucinolone Acetonide Intraocular Implant | Standard Systemic Treatment
Started | 129 (129 participants were assigned to implant; 122 received implant) | 126 (126 participants were assigned to systemic treatment; 121 received systemic therapy)
Completed | 118 (118 participants completed the 2-year anniversary visit) | 114 (114 participants completed the 2-year anniversary visit)
Not Completed | 11 | 12
Not completed — Lost to Follow-up | 5 | 8
Not completed — Missed 2-year visit | 4 | 4
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flucinolone Acetonide Intraocular Implant | Standard Systemic Treatment | Total
Number analyzed (Participants) | 129 | 126 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (15) | 47 (15) | 46 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 100 | 191
  Male | 38 | 26 | 64
Race/Ethnicity, Customized [Number; unit: participants]
  White | 72 | 70 | 142
  Hispanic | 18 | 15 | 33
  Black | 35 | 31 | 66
  Other | 4 | 10 | 14
Region of Enrollment [Number; unit: participants]
  United States | 109 | 104 | 213
  Australia | 5 | 6 | 11
  United Kingdom | 15 | 16 | 31
Bilateral uveitis [Number; unit: participants] | 116 | 108 | 224
Site of uveitis [Number; unit: participants]
  Intermediate | 50 | 47 | 97
  Posterior or Panuveitis | 79 | 79 | 158
Associated systemic inflammatory disease [Number; unit: participants]
  Yes | 36 | 33 | 69
  no | 93 | 93 | 186
Visual acuity 20/40 or better [Number; unit: eyes] | 116 | 122 | 238
Active uveitis [Number; unit: eyes] | 192 | 181 | 373
Visual acuity 20/200 or worse [Number; unit: eyes] | 39 | 35 | 74

OUTCOME MEASURES:

1. Primary Outcome: Change in Best-corrected Visual Acuity (Change in the Numbers of Letters Read From a Standard ETDRS Eye Chart) From Baseline to 24 Months in Eyes With Uveitis
Description: Best-corrected visual acuity was measured as the number of letters read from standard logarithmic visual acuity charts by study-certified examiners who were masked to treatment. Visual acuity was measured at all study visits. The primary outcome was eye-specific change in visual acuity from baseline to 2-year follow-up. Positive change values indicate improved vision while negative change values indicate vision has gotten worse. A change of 7.5 letters is considered clinically meaningful.
Time Frame: 24 months
Population: The primary analysis was an intention-to-treat analysis; analysis was conducted "as randomized". Data from the 255 randomized participants were used in the analytic model. 232 of the 255 completed the 2 year outcome visit.
Measure: Mean (Standard Error); unit: letters
Groups:
- Flucinolone Acetonide Implant: A fluocinolone acetonide intravitreal implant (0.59 mg) was surgically placed by a study-certified surgeon was placed in each eligible eye. The first eye was implanted within 28 days of randomization and, if eligible, the second eye within the next 28 days. Prior to implant surgery, topical, periocular or systemic corticosteroids where used as needed to quiet the anterior chamber. Post-implant, systemic corticosteroids and immunosuppressive drugs were tapered and discontinued. If the second eye was not eligible for an implant initially but later became eligible, an implant was placed in the second eye at that time. The treatment algorithm included re-implantation upon reactivation and treatment per best medical judgment for failure to achieve inflammation control, treatment-limiting toxicity and systemic disease requiring systemic therapy.
- Systemic Therapy: Oral corticosteroids supplemented with immunosuppressive drugs if indicated were given according to published guidelines developed by an expert panel. For participants with active uveitis at baseline, 1 mg/kg/day up to 60 mg/day of prednisone was given until uveitis was controlled or 4 weeks had elapsed. When control was achieved, prednisone was tapered per study guidelines. Immunosuppressive drugs were added when uveitis was not initially controlled with prednisone alone, as corticosteroid-sparing agents when prednisone could not be tapered to 10 mg/day without reactivation of uveitis and for specific uveitis syndromes. Choice of immunosuppressant was made by the study ophthalmologist; immunosuppressant administration and monitoring for toxicity was conducted according to expert guidelines.
Arm/Group | Flucinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 129 | 126
letters | 6.0 (1.4) | 3.2 (1.4)
Statistical Analysis 1: Comparison: Flucinolone Acetonide Implant vs Systemic Therapy; Null hypothesis: There will be no difference in change in visual acuity between treatment groups. Assuming 67% bilateral disease, between eye correlation of 0.4, SD of 16 letters' change over 2 years and two-sided type 1 error rate of .05, a sample size of 250 provided 91% power (assuming 10% crossover) to detect a treatment difference of 7.5 standard ETDRS letters' change in visual acuity from baseline to 24 months; Test type: Superiority or Other; p = 0.16, Generalized estimating equations, linear — unadjusted; Mean Difference (Net) = 2.79, 95% CI 2-sided [-1.16 to 6.68], Standard Error of Mean 2.03 — The treatment effect is a model-based comparison of within group treatment change from enrollment to 24 months (the difference of the differences - implant minus systemic)

2. Secondary Outcome: Macular Edema
Description: center point macular thickness >= 240 micrometers assessed on OCT (Stratus OCT-3 [Carl Zeiss Meditec, Dublin, CA]) as graded by Central Reading Center
Time Frame: 24 months
Population: All eyes with uveitis were included in the analysis (245 eyes of the 129 participants randomized to implant therapy and 234 eyes of the 126 participants randomized to systemic therapy)..
Measure: Number (95% Confidence Interval); unit: percentage of eyes with uveitis
Units Other Than Participants: eyes with macular edema
Groups:
- Flucinolone Acetonide Implant: Participants randomized to receive implant therapy.
- Systemic Therapy: Participants randomized to receive systemic therapy.
Arm/Group | Flucinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 129 | 126
Number analyzed (eyes with macular edema) | 245 | 234
percentage of eyes with uveitis | 22 [14 to 30] | 30 [21 to 40]
Statistical Analysis 1: Comparison: Flucinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p = 0.071, GEE, logistic — unadjusted; Ratio of odds ratios = 0.61, 95% CI 2-sided [0.34 to 1.03] — For each treatment group the odds of macular edema at 2 yrs as compared to baseline was computed. The treatment effect is the ratio of these odds (implant divided by systemic)

3. Secondary Outcome: Uveitis Activity
Description: Uveitis activity was determined by clinician assessment at each study visit. The study ophthalmologist evaluated each eye as active, inactive/never had uveitis or cannot assess.
Time Frame: 24 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of eyes with uveitis
Units Other Than Participants: eyes with uveitis
Groups:
- Fluocinolone Acetonide Implant: Participants randomized to receive implant therapy
Arm/Group | Fluocinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 129 | 126
Number analyzed (eyes with uveitis) | 245 | 234
percentage of eyes with uveitis | 12 [06 to 20] | 29 [21 to 39]
Statistical Analysis 1: Comparison: Fluocinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p = 0.001, GEE, logistic — unadjusted; Ratio of odds ratios = .29, 95% CI 2-sided [.13 to .60] — For each treatment group the odds of uveitis activity at 2 years as compared to baseline was computed. The treatment effect represents the ratio of these odds (implant divided by systemic)

4. Secondary Outcome: Intraocular Pressure - Incident IOP Greater Than or Equal to 30 mm Hg
Time Frame: 24 months
Population: Eyes, not participants, were analyzed. Eyes with prevalent complications or missing data at enrollment were were excluded from the risk set.
Measure: Number (95% Confidence Interval); unit: percentage of eyes with uveitis at risk
Units Other Than Participants: eyes with uveitis
Arm/Group | Flucinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 129 | 126
Number analyzed (eyes with uveitis) | 234 | 229
percentage of eyes with uveitis at risk | 32.8 [27.1 to 39.2] | 6.3 [3.7 to 10.3]
Statistical Analysis 1: Comparison: Flucinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p < .0001, Cox proportional hazards w/ RE — unadjusted; Hazard Ratio (HR) = 6.08, 95% CI 2-sided [3.32 to 11.15] — A Cox proportional hazards model with a random effect to account for between-eye correlation was used to estimate the relative hazard of experiencing an IOP of 30 mmHg or greater. The systemic arm was the reference group

5. Secondary Outcome: Intraocular Pressure - Incident IOP Greater Than or Equal to 24 mm Hg
Time Frame: 24 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of eyes with uveitis at risk
Units Other Than Participants: eyes with uveitis
Arm/Group | Flucinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 129 | 126
Number analyzed (eyes with uveitis) | 234 | 228
percentage of eyes with uveitis at risk | 53.1 [46.9 to 59.7] | 18.7 [14.2 to 24.5]
Statistical Analysis 1: Comparison: Flucinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p < .0001, Cox proportional hazards w/ RE — unadjusted; Hazard Ratio (HR) = 3.59, 95% CI 2-sided [2.34 to 5.50] — A Cox proportional hazards model with a random effect to account for between-eye correlation was used to estimate the relative hazard of experiencing an IOP of 24 mmHg or greater. The systemic arm was the reference group

6. Secondary Outcome: Intraocular Pressure - Incident IOP Elevation >= 10 mmHg Above Baseline
Time Frame: 24 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of eyes with uveitis at risk
Units Other Than Participants: eyes with uveitis
Arm/Group | Fluocinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 129 | 126
Number analyzed (eyes with uveitis) | 235 | 230
percentage of eyes with uveitis at risk | 51.8 [45.5 to 58.3] | 15.5 [11.4 to 20.9]
Statistical Analysis 1: Comparison: Fluocinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p < .0001, Cox proportional hazards with RE — unadjusted; Hazard Ratio (HR) = 4.28, 95% CI 2-sided [2.78 to 6.58] — A Cox proportional hazards model with a random effect to account for between-eye correlation was used to estimate the relative hazard of experiencing an IOP that was 10mmHg or greater than the baseline value. The systemic arm was the reference group

7. Secondary Outcome: Glaucoma - Incident
Description: Glaucoma was diagnosed by a glaucoma specialist through review of visual fields, clinical data, and fundus images.
Time Frame: 24 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of eyes with uveitis at risk
Units Other Than Participants: eyes with uveitis
Arm/Group | Fluocinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 129 | 126
Number analyzed (eyes with uveitis) | 212 | 202
percentage of eyes with uveitis at risk | 16.5 [12.1 to 22.2] | 4.0 [2.0 to 7.8]
Statistical Analysis 1: Comparison: Fluocinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p = 0.0008, Cox proportional hazards w/ RE — unadjusted; Hazard Ratio (HR) = 4.19, 95% CI 2-sided [1.82 to 9.63] — A Cox proportional hazards model with a random effect to account for between-eye correlation was used to estimate the relative hazard of developing glaucoma. The systemic arm was the reference group

8. Secondary Outcome: Intraocular Pressure (IOP) - Incident Use of IOP-lowering Medical Therapy (Percentage of Eyes With Uveitis That Were Not Being Treated With IOP-lowering Medical Therapy at Baseline and Underwent IOP Lowering Therapy During the 24 Month Follow-up.
Description: The percentage of subjects who used topical or systemic treatment for elevated IOP at any time during the 2 year follow-up and were not on IOP-lowering therapy at baseline is reported.
Time Frame: 24 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of eyes with uveitis at risk
Units Other Than Participants: eyes
Arm/Group | Flucinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 129 | 126
Number analyzed (eyes) | 201 | 203
percentage of eyes with uveitis at risk | 61.1 [54.3 to 67.8] | 20.1 [15.1 to 26.3]
Statistical Analysis 1: Comparison: Flucinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p < .0001, Cox proportional hazards w/ RE — unadjusted; Hazard Ratio (HR) = 4.16, 95% CI 2-sided [2.67 to 6.47] — A Cox proportional hazards model with a random effect to account for between-eye correlation was used to estimate the relative hazard of using an IOP-lowering therapy. The systemic arm was the reference group

9. Secondary Outcome: Intraocular Pressure - IOP-lowering Surgery
Time Frame: 24 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of eyes with uveitis at risk
Units Other Than Participants: eyes with uveitis
Arm/Group | Flucinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 129 | 126
Number analyzed (eyes with uveitis) | 233 | 226
percentage of eyes with uveitis at risk | 26.2 [21.0 to 32.4] | 3.7 [1.9 to 7.2]
Statistical Analysis 1: Comparison: Flucinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p < 0.0001, Cox proportional hazards w/ RE — unadjusted; Hazard Ratio (HR) = 8.40, 95% CI 2-sided [3.39 to 20.82] — A Cox proportional hazards model with a random effect to account for between-eye correlation was used to estimate the relative hazard of having surgery to lower IOP. The systemic arm was the reference group

10. Secondary Outcome: Cataract - Incident Cataract
Time Frame: 24 months
Population: Eyes with uveitis, not participants, were analyzed. Eyes with prevalent complications or missing data at enrollment were were excluded from the risk set.
Measure: Number (95% Confidence Interval); unit: percentage of eyes with uveitis at risk
Units Other Than Participants: eyes with uveitis
Arm/Group | Fluocinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 129 | 126
Number analyzed (eyes with uveitis) | 54 | 50
percentage of eyes with uveitis at risk | 90.7 [81.3 to 96.6] | 44.9 [32.3 to 59.8]
Statistical Analysis 1: Comparison: Fluocinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p < 0.0001, Cox proportional hazards w/ RE — unadjusted; Hazard Ratio (HR) = 4.12, 95% CI 2-sided [2.21 to 7.67] — A Cox proportional hazards model with a random effect to account for between-eye correlation was used to estimate the relative hazard of developing a cataract. The systemic arm was the reference group

11. Secondary Outcome: Change in Self-reported Vision-related Function as Measured by the National Eye Institute 25-Item Visual Function Questionnaire (NEI-VFQ 25) Vision Targeted Composite Score From Baseline to 24 Months
Description: The NEI-VFQ 25 measures the effect of visual disability/symptoms with generic health and task-oriented domains. The range for the composite score is 0 to 100; higher scores are associated with better visual function. A change of 4 to 6 points is considered to be a clinically meaningful difference.
Time Frame: 24 months
Measure: Mean (Standard Error); unit: units on a scale (composite score)
Arm/Group | Fluocinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 129 | 126
units on a scale (composite score) | 11.44 (1.67) | 6.80 (1.58)
Statistical Analysis 1: Comparison: Fluocinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p = 0.043, GEE, linear — unadjusted; Mean Difference (Net) = 4.64, 95% CI 2-sided [0.14 to 9.15], Standard Error of Mean 2.30 — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Change in SF-36 Mental Component Score From Baseline to 24 Months
Description: Self-reported health related QoL was measured with the SF 36 survey. The mental component score for the SF 36 is a summary measure of mental health primarily based on the social functioning, role emotional, mental health and vitality domains. The score is scaled to a population norm with a mean of 50 and standard deviation of 10. Higher scores represent better outcomes. The mean change in scores between baseline and 24 months was calculated for each treatment group.
Time Frame: 24 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Flucinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 129 | 126
units on a scale | 2.55 (1.11) | -1.1 (1.15)
Statistical Analysis 1: Comparison: Flucinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p = 0.023, GEE, linear — unadjusted; Mean Difference (Net) = 3.62, 95% CI 2-sided [0.49 to 6.76], Standard Error of Mean 1.60 — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Change in SF-36 Physical Component Score From Baseline to 24 Months
Description: Self-reported health related QoL was measured with the SF 36 survey. The physical component score for the SF 36 is a summary measure of physical health primarily based on the physical functioning, role physical, bodily pain and general health domains of the survey. The score is scaled to a population norm with a mean of 50 and standard deviation of 10. Higher scores represent better outcomes. The mean change in scores between baseline and 24 months was calculated for each treatment group. A 3 to 5 point difference is considered to be clinically meaningful.
Time Frame: 24 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Flucinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 129 | 126
units on a scale | 1.15 (0.83) | -1.8 (0.90)
Statistical Analysis 1: Comparison: Flucinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p = 0.016, Generalized Estimating Equations — unadjusted; Mean Difference (Net) = 2.95, 95% CI 2-sided [0.54 to 5.36], Standard Error of Mean 1.23 — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Hyperlipidemia - Incident
Description: LDL greater than or equal to 160 mg/mL
Time Frame: 24 months
Population: Number of participants at risk were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants at risk
Arm/Group | Flucinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 97 | 104
percentage of participants at risk | 9.8 [5.2 to 18.0] | 11.0 [6.3 to 19.1]
Statistical Analysis 1: Comparison: Flucinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p = 0.84, Regression, Cox — unadjusted; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.39 to 2.15] — A Cox proportional hazards model was used to evaluate the relative hazard of hyperlipidemia for the implant and systemic treatments. The systemic treatment is the reference group

15. Secondary Outcome: Hypertension Diagnosis Requiring Treatment
Time Frame: 24 months
Population: Participants with prevalent complications or missing data at enrollment were excluded from the risk set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Flucinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 88 | 88
percentage of participants | 4.6 [1.8 to 11.9] | 10.5 [5.6 to 19.3]
Statistical Analysis 1: Comparison: Flucinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p = 0.13, Regression, Cox — unadjusted; Hazard Ratio (HR) = 0.40, 95% CI 2-sided [0.13 to 1.29] — A Cox proportional hazards model was used to evaluate the relative hazard of hypertension for the implant and systemic treatments. The systemic treatment is the reference group

16. Secondary Outcome: Diabetes Mellitus
Time Frame: 24 months
Population: Participants with prevalent complications or missing data at enrollment were excluded from the risk set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Flucinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 105 | 114
percentage of participants | 1.0 [0.1 to 6.6] | 3.6 [1.4 to 9.4]
Statistical Analysis 1: Comparison: Flucinolone Acetonide Implant vs Systemic Therapy; Test type: Superiority or Other; p = 0.24, Regression, Cox — unadjusted; Hazard Ratio (HR) = 0.26, 95% CI 2-sided [0.03 to 2.44] — A Cox proportional hazards model was used to evaluate the relative hazard of diabetes mellitus for the implant and systemic treatments. The systemic treatment is the reference group

17. Secondary Outcome: Mortality
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Flucinolone Acetonide Implant | Systemic Therapy
Number analyzed (Participants) | 126 | 124
percentage of participants | 1.6 [0.4 to 6.3] | 0 [NA to NA] — no deaths reported in systemic group

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Flucinolone Acetonide Implant | Systemic Therapy
Serious Adverse Events (participants affected / at risk) | 75/129 | 47/126
Other Adverse Events (participants affected / at risk) | 113/129 | 113/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Flucinolone Acetonide Implant (N=129) | Systemic Therapy (N=126)
Endophthalmitis (Eye disorders) | 3 (3) | 0 (0)
Glaucoma (Eye disorders) | 7 (11) | 1 (2)
Hypotony (Eye disorders) | 4 (4) | 2 (2)
Ocular Hypertension (Eye disorders) | 32 (54) | 5 (6)
Retinal Detachment (Eye disorders) | 4 (5) | 1 (1)
Vitreous Hemorrhage (Eye disorders) | 14 (15) | 4 (5)
Bleb revision (Eye disorders) | 1 (1) | 0 (0)
Complication of Kenalog injection (Eye disorders) | 1 (1) | 0 (0)
Enucleation (Eye disorders) | 0 (0) | 1 (1)
Hospitalization for cataract surgery (Eye disorders) | 0 (0) | 1 (2)
Retisert wound dehiscence (Eye disorders) | 1 (1) | 0 (0)
Choroidal neovascularization (Eye disorders) | 1 (1) | 0 (0)
Hyphema (Eye disorders) | 1 (1) | 0 (0)
Exposed suture (Eye disorders) | 1 (1) | 0 (0)
Surgery to reposition shunt (Eye disorders) | 1 (1) | 0 (0)
Iris bombe (Eye disorders) | 1 (1) | 0 (0)
Exposed Ahmed valve (Eye disorders) | 1 (1) | 0 (0)
Orbital cellulitis (Eye disorders) | 1 (1) | 0 (0)
Revision of Ahmed valve (Eye disorders) | 1 (1) | 0 (0)
Abnormal ERG (Eye disorders) | 0/120 (0) | 1 (1)
Hospitalization for observation while on prednisone (Psychiatric disorders) | 1 (1) | 0 (0)
Anterior cervical dissection, fusion (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhea, dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileostomy takedown (Gastrointestinal disorders) | 0 (0) | 1 (1)
Perforated viscus lung cancer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pericardial drain placement (Cardiac disorders) | 0 (0) | 1 (1)
Hysterectomy (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Kidney stones (Renal and urinary disorders) | 1 (1) | 0 (0)
Hip replacement (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Precancerous cells right breast (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prolonged hospitalization stay due to reaction (General disorders) | 1/120 (1) | 0 (0)
Shoulder surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Total thyroidectomy (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (General disorders) | 0 (0) | 1 (1)
Arthrosis due to aseptic necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dislocation of hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exacerbation of intestinal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flu-like reaction to Avonex (General disorders) | 0 (0) | 1 (1)
Gall bladder surgery (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hypertension (Cardiac disorders) | 7 (12) | 3 (5)
Hemmorhagic cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hospitalization (General disorders) | 0 (0) | 1 (1)
Hospitalization for post-surgical observation of pharyngeal papilloma biopsy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Torn medial meniscus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neuro Bechet's disease (Immune system disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Psychotic episode (Psychiatric disorders) | 0 (0) | 1 (1)
Abnormal laboratory value (Hepatobiliary disorders) | 4 (5) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Infection (Infections and infestations) | 6 (9) | 5 (5)
Miscarriage (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Non-melanoma skin cancer (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (7)
Cardiovascular (Cardiac disorders) | 2 (2) | 4 (5)
Thrombosis (Vascular disorders) | 4 (4) | 2 (2)
Headache due to hypertension (General disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
Chest pain (Investigations) | 1 (2) | 3 (3)
Gastrointestinal (Gastrointestinal disorders) | 1 (3) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flucinolone Acetonide Implant (N=129) | Systemic Therapy (N=126)
Hyperglycemia (fasting) (Metabolism and nutrition disorders) | 4 (4) | 10 (16)
Hyperglycemia (casual) (Metabolism and nutrition disorders) | 6 (8) | 10 (16)
Hypoglycemia (Metabolism and nutrition disorders) | 7 (8) | 6 (6)
Triglyceride (high) (Metabolism and nutrition disorders) | 10 (12) | 10 (12)
SGOT (AST) or SGPT (ALT) (Hepatobiliary disorders) | 5 (9) | 8 (13)
BUN (Renal and urinary disorders) | 8 (8) | 10 (16)
Nausea (Gastrointestinal disorders) | 5 (7) | 20 (24)
Vomiting (Gastrointestinal disorders) | 5 (5) | 11 (15)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 12 (16)
Mood (Psychiatric disorders) | 4 (4) | 11 (12)
Headache (General disorders) | 25 (36) | 19 (21)
Fatigue (General disorders) | 6 (7) | 11 (15)
Hypertension (systolic) (Cardiac disorders) | 27 (38) | 32 (62)
Hypertension (diastolic) (Cardiac disorders) | 24 (39) | 30 (47)
Allergic reaction (Immune system disorders) | 10 (16) | 9 (11)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 12 (12) | 10 (10)
Infection (General disorders) | 52 (116) | 67 (178)
Ocular hypertension (Eye disorders) | 78 (246) | 29 (67)
Glaucoma (Eye disorders) | 10 (13) | 2 (5)
Hypotony (Eye disorders) | 26 (46) | 10 (28)
Cataract (Eye disorders) | 40 (65) | 13 (15)
Vitreous hemorrhage (Eye disorders) | 13 (15) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No